CLINICAL TRIAL: NCT01617447
Title: A Short-term Administration Study of Aripiprazole in Children and Adolescents (Age: 6 to 17 Years) With Autistic Disorder
Brief Title: A Short Treatment Study of Aripiprazole in Pediatric Patients With Autistic Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 031-11-002
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-02

CONDITIONS: Autistic Disorder
Keywords: Autistic Disorder, children and adolescents; Aripiprazole; Double-blind; Randomized; children and adolescents
MeSH Terms: conditions — Autistic Disorder | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): administered orally once daily
  Interventions: Drug: Placebo of Aripiprazole
- Aripiprazole (Experimental): administered orally once daily
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Placebo of Aripiprazole — administered orally once daily
  Arms: Placebo
Drug: Aripiprazole — Flexibly dose administered orally once daily
  Arms: Aripiprazole

SUMMARY:
The objective of this study is to investigate the efficacy and safety of aripiprazole orally administered over a period of 8 weeks in pediatric patients with Autistic Disorder

ELIGIBILITY:
Inclusion Criteria:

* The patient meets current DSM-IV-TR diagnostic criteria for Autistic Disorder (defined in DSM-IV-TR) and also demonstrates behaviors such as tantrums, aggression, self-injurious behavior, or a combination of these problems.
* Inpatient or outpatient status
* Others

Exclusion Criteria:

* The patient is currently diagnosed with another disorder on the autism spectrum in DSM-IV-TR, including Asperger's, Rett's Disorder, PDD-NOS, Childhood Disintegrative Disorder, or Fragile-X Syndrome.
* Patients who fall under a contraindication listed in the ABILIFY package insert
* Others

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2012-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyoji Imaoka, Mr, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (5):
- Japan (5):
  - Chubu Region
  - Chugoku Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711

RESULTS

PARTICIPANT FLOW:
Groups:
- Aripiprazole: Aripiprazole were orally administered once daily for 8 weeks. The starting dose was 1 mg/day, and the dose will be escalated to 3, 6, 9, 12, and 15 mg/day in a stepwise manner. The dose was fixed after Week 6 and administration continued for another 2 weeks until Week 8.
- Placebo: Placebo were orally administered once daily for 8 weeks.
Period: Overall Study
Arm/Group | Aripiprazole | Placebo
Started | 47 | 45
Completed | 47 | 42
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole | Placebo | Total
Number analyzed (Participants) | 47 | 45 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 47 | 45 | 92
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.3 (3.3) | 9.9 (3.1) | 10.1 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 39 | 36 | 75
Region of Enrollment [Number; unit: participants]
  Japan | 47 | 45 | 92

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Aberrant Behavior Checklist Japanese Version (ABC-J) Irritability Subscale Score
Description: The ABC-J Irritability subscale consists of 15 items. Each item scores range from 0 to 3: 0 = No problem, 1 = Mild aberrant behavior, 2 = Moderate aberrant behavior, and 3 = Severe aberrant behavior. Individual scores were summed, therefore, the overall score range was between 0-45. Higher scores represent worse condition.
Time Frame: baseline, 8 weeks after dosing
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 47 | 45
units on a scale | -11.4 (1.3) | -7.5 (1.4)

ADVERSE EVENTS:
Time Frame: From the start date of investigational medicinal product (IMP) administration to date of the final examination (up to Week 8 at e hours after IMP administration)
Arm/Group | Aripiprazole | Placebo
Serious Adverse Events (participants affected / at risk) | 0/47 | 1/45
Other Adverse Events (participants affected / at risk) | 39/47 | 32/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (N=47) | Placebo (N=45)
Heat illness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (N=47) | Placebo (N=45)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Malaise (General disorders) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 4 (4)
Nasopharyngitis (Infections and infestations) | 10 (18) | 11 (12)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (6)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 1 (1)
Somnolence (Nervous system disorders) | 24 (25) | 4 (4)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 2 (2) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Perianal erythema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Decreased activity (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Local swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Thirst (General disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (2)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (4) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1)
Hyperphagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Akathisia (Nervous system disorders) | 1 (1) | 0 (0)
Autism (Nervous system disorders) | 0 (0) | 1 (1)
Bradykinesia (Nervous system disorders) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 0 (0)
Sedation (Nervous system disorders) | 1 (1) | 0 (0)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Apathy (Psychiatric disorders) | 1 (1) | 0 (0)
Emotional disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Parasomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Self injurious behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4)
Laryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No